CLINICAL TRIAL: NCT05183464
Title: Analysis of New Salivary Biomarkers to Evaluate Excessive Diurnal Sleepiness in Children With Hypersomnia
Acronym: BIOSOM
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_1119; 2021-A02740-41 (Other: ID-RCB)
Record Dates: First submitted 2021-12-21; First posted 2022-01-10 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Hypersomnia; Sleepiness, Excessive Daytime
Keywords: Excessive Diurnal Sleepiness; Salivary biomarkers; Children, a-amylase; oxalate; Hypersomnia; sleep
MeSH Terms: conditions — Disorders of Excessive Somnolence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Children with primary hypersomnia: Children with primary hypersomnia, i.e. narcolepsy or idiopathic hypersomnia
  Interventions: Biological: saliva samples; Behavioral: Stanford sleepiness scale; Behavioral: Karolinska Sleepiness Scale; Behavioral: Epworth Sleepiness Scale; Behavioral: BLAST test
- Children with secondary hypersomnia: Children with a secondary hypersomnia, i.e. caused by sleep deprivation, a psychiatric disorder, sleep fragmentation, circadian delay.
  Interventions: Biological: saliva samples; Behavioral: Stanford sleepiness scale; Behavioral: Karolinska Sleepiness Scale; Behavioral: Epworth Sleepiness Scale; Behavioral: BLAST test

INTERVENTIONS:
Biological: saliva samples — Collection of salivary a-amylase during the day (5 times a day: at 8:00 am, 9:00 am,1:00pm, 4:00pm and 8:00pm) with Salivette.
Behavioral: Stanford sleepiness scale — The Stanford Sleepiness Scale evaluates sleepiness at the time of the evaluation. The subjects have to choose the statement best representing their level of sleepiness on a scale ranging from 1 to 7: the higher the score, the higher the sleepiness.
  This scale will be submitted to the children before each salivary sampling (5 times a day: at 8:00 am, 9:00 am,1:00pm, 4:00pm and 8:00pm)
Behavioral: Karolinska Sleepiness Scale — The Karolinska Sleepiness Scale assesses the perceived level of sleepiness at the time of the evaluation on a 9-points scale. The higher the score, the higher the sleepiness.
  This scale will be submitted to the children before each salivary sampling (5 times a day: at 8:00 am, 9:00 am,1:00pm, 4:00pm and 8:00pm)
Behavioral: Epworth Sleepiness Scale — The Adapted Epworth Sleepiness Scale for children in which the item "falling asleep while in a car stopped in traffic" was replaced by "falling asleep at school" assesses the risk of falling asleep in 8 daily-life situations estimated on a 4-point Likert scale. The total score is the sum of the scores for the 8 items: a higher score represents greater sleepiness and the pathological threshold is higher than 10.
  This scale will be submitted to the children one time, at the onset of the hospitalization.
Behavioral: BLAST test — The BLAST (Bron/Lyon Attention Stability Test) is a computerized attention test evaluating brief lapses of attention with 4 measures: reaction times, errors and two composite measures (Stability and Intensity). The subjects have to detect the presence or the absence of a specific stimulus during approximatively 60 trials for 3 minutes. Normative data are available for both children and adults.
  This test is part of the neuropsychological evaluation, conducted the afternoon of the first day of hospitalization. The test is realized at 4:00pm.

SUMMARY:
Excessive diurnal sleepiness is characterized by an incapacity to stay awake, in favour of sleep occurrence. This sleepiness might be secondary to a sleep disorder; when it is not the case, it is primary hypersomnia (including narcolepsy and idiopathic hypersomnia).

To date, objective measures of sleepiness can only be achieved in laboratory. Subjective techniques as scales and questionnaires are highly sensitive to inter-individual differences and cannot constitute a reliable diagnosis tool of sleepiness.

Recent studies suggested that some salivary biomarkers are sensitive to sleep characteristics and thus, may allow the objective and easy evaluation of sleepiness.

The objective of the study is to explore the usability of salivary biomarkers (a-amylase and oxalate) as a new non-invasive technique to evaluate sleepiness and to diagnose primary hypersomnia in children.

The hypothesis of this study is that there will be a modification of salivary biomarkers concentrations with the variations of diurnal sleepiness.

ELIGIBILITY:
Inclusion Criteria:

* Children with excessive diurnal sleepiness hospitalized for an evaluation of hypersomnia symptoms
* Age> 6 years old and <18 years old
* Non opposition by both parents

Exclusion Criteria:

* Opposition of the child or parents to participate
* Patients under measure of deprivation of rights and liberty

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children hospitalized for an evaluation of their excessive diurnal sleepiness will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Salivary a-amylase concentration (U/ml) | 3 days following the inclusion
  Salivary a-amylase concentrations will be collected with Salivette. Children will be asked to passively keep a piece of cotton in mouth that will absorb the saliva for one minute.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Mère-Enfant - Service d'épileptologie clinique, des troubles du sommeil et de neurologie fonctionnelle de l'enfant, Bron, France